CLINICAL TRIAL: NCT01003041
Title: The Influence of Hearing Discrete Phonemes in Mother's Voice in the Infant's Natural Environment and With Natural Melody on Developing Phonetic Categories Between 4-10 Months Old
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maaynei Hayesha Medical Center (Other)
Responsible Party: DR OPHIR, maaynei hayeshoa
Other Study IDs: 1010
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2009-10-28 (Estimated); Status verified 2009-10

CONDITIONS: Healthy
Keywords: healthy normal infants

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

GROUPS / COHORTS (1):
- lifestyle counseling: in the future parents will be advised to expose their infants to phonetic sounds in order to develop their phonetic categories in the future

SUMMARY:
The purpose of this study is to record voice samples of infant's mothers, process in samples to a phonetic musical piece, play the phonetic musical piece to 4-10 month old infants, and then test the infants in a conditioned head turning test in lab, and to analyze the results.

ELIGIBILITY:
Inclusion Criteria:

* normal newborn infants
* males and females
* age 4 months to 10 months old

Exclusion Criteria:

* chronic illness
* hearing loss
* history of otitis media
* serious otitis media

Ages: 4 Months to 10 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: normal newborn infants
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-10

PRIMARY OUTCOMES:
Response by head-turning test to familiar and unfamiliar phonetic categories | one year